CLINICAL TRIAL: NCT01326429
Title: Frequency and Origin of Dysnatremias in the Emergency Department
Status: Withdrawn | Type: Observational
Why Stopped: Job change of responsible investigators
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Steering committee of the NCCR (Unknown)
Responsible Party: Gregor Lindner M.D., Dept. of Nephrology and Hypertension, Inselspital Bern, University of Bern
Other Study IDs: KEK 019/11
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Hyponatremia; Hypernatremia
Keywords: Sodium; Hyponatremia; Hypernatremia; Emergency department
MeSH Terms: conditions — Hyponatremia; Hypernatremia; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypernatremia: Patients admitted to the emergency department with a serum sodium exceeding 145 mmol/L.
- Hyponatremia: Patients admitted to the emergency room with a serum sodium below 135 mmol/L.

SUMMARY:
Hypo- and hypernatremia are the most frequent electrolyte disorders found in hospitalized patients. The increasing use of diuretics and other medications influencing the water and sodium homeostasis potentially lead to a rise in the prevalence of the electrolyte disorders. Only little data is available on the frequency and the mechanisms leading to hypo-/hypernatremia.

Thus, the investigators aim to A.) determine the frequency of hypo- and hypernatremia in the emergency department of a large tertiary university hospital and B.) explore the mechanisms leading to the development of dysnatremias by detailed clinical and laboratory examinations.

ELIGIBILITY:
Inclusion Criteria:

* Serum sodium below 135 mmol/L (i.e. hyponatremia); serum sodium exceeding 145 mmol/L (hypernatremia)

Exclusion Criteria:

* Patients below age 18 years; patients declining study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the emergency department of a large tertiary university hospital with a serum sodium below 135 mmol/L (hyponatremia) or exceeding 145 mmol/L.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Frequency of hypo- and hypernatremia in the emergency department | approx. 6 months
  The investigators aim to determine the frequency of hypo- and hypernatremia in the emergency department of a large tertiary university hospital.

SECONDARY OUTCOMES:
Origin of hypo- and hypernatremia in the emergency department | approx. 6 months
  The investigators try to investigate the mechanisms leading to the development of hypo- and hypernatremia in patients admitted to the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Lindner, M.D., Principal Investigator — Dept. of Nephrology and Hypertension, Inselspital Bern, University of Bern; Felix J Frey, M.D., Study Chair — Dept. of Nephrology and Hypertension, Inselspital Bern, University of Bern

REFERENCES:
- See also: Institution homepage — http://nephrologie.insel.ch